CLINICAL TRIAL: NCT05129891
Title: A Study Investigating Pharmacokinetic Properties When Dosing Different Formulations of Oral Peptide Therapeutics in Healthy Male Participants
Brief Title: A Research Study Looking at New Protein-based Tablets in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9501-4821; U1111-1266-0672 (Other: World Health Organization (WHO)); 2021-001452-34 (EudraCT Number)
Record Dates: First submitted 2021-08-09; First posted 2021-11-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers; High Blood Cholesterol Levels; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: Oral semaglutide (Experimental): Four different formulations of oral semaglutide are investigated. One formulation given for 10 days before participants receive a different formulation for 5 days
  Interventions: Drug: Semaglutide D; Drug: Semaglutide G; Drug: Semaglutide H; Drug: Semaglutide I
- Part B: NNC0385-0434 (Experimental): Four different formulations of NNC0385-0434 are investigated. One formulation given for 10 days before participants receive a different formulation for 5 days
  Interventions: Drug: NNC0385-0434 B; Drug: NNC0385-0434 C; Drug: NNC0385-0434 D; Drug: NNC0385-0434 E

INTERVENTIONS:
Drug: Semaglutide D — Tablet given orally
  Arms: Part A: Oral semaglutide
Drug: Semaglutide G — Tablet given orally
  Arms: Part A: Oral semaglutide
Drug: Semaglutide H — Tablet given orally
  Arms: Part A: Oral semaglutide
Drug: Semaglutide I — Tablet given orally
  Arms: Part A: Oral semaglutide
Drug: NNC0385-0434 B — Tablet given orally
  Arms: Part B: NNC0385-0434
Drug: NNC0385-0434 C — Tablet given orally
  Arms: Part B: NNC0385-0434
Drug: NNC0385-0434 D — Tablet given orally
  Arms: Part B: NNC0385-0434
Drug: NNC0385-0434 E — Tablet given orally
  Arms: Part B: NNC0385-0434

SUMMARY:
In this study, four new tablet versions of two compounds will be investigated.

The aim of this study is to investigate the amount of the active ingredient and helping agent in the blood after doses of four different tablet versions. The tablet versions, participants will receive, i.e. the treatment arm participants will be assigned to, is decided by chance.

Participants will receive one treatment for 10 days in the first period. For the second period, directly following, participants will receive a different treatment for five more days.

The study can last for up to approximately 10 weeks for each participant. This includes a screening period (up to 3 weeks), two treatment periods (together a total of 15 days) and a follow-up visit (5 weeks after the last dosing)

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index between 20.0 and 29.9 kg/m^2 (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to study interventions or related products.
* Use of prescription medicinal products or non-prescription drugs (including herbal products and vaccines), except routine vitamins and topical medications not reaching the systemic circulation, within 14 days prior to the day of screening.
* Any disorder which in the investigator's opinion might jeopardise participant safety or compliance with the protocol.
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator.
* History (as declared by the participant or reported in the medical records) of major surgical procedures involving the stomach potentially affecting absorption of study products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 384 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,API,day10; area under the API plasma concentration-time curve from 0 to 24 hours after the 10th dose | From pre-dose PK sample (0 hours) at day 10 to PK sample 24 hours after dose administration
  h * nmol/L

SECONDARY OUTCOMES:
Cmax,API,day10; maximum observed plasma concentration of API after the 10th dose | From pre-dose PK sample (0 hours) at day 10 to PK sample 24 hours after dose administration
  nmol/L
tmax, API,day10; time from the 10th dose to maximal observed plasma concentration of API | From pre-dose PK sample (0 hours) at day 10 to PK sample 24 hours after dose administration
  hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Altasciences Company Inc., Montreal, Quebec, Canada
- Parexel International GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com